CLINICAL TRIAL: NCT01576952
Title: A Randomized Double-Masked Study to Compare the Ocular Safety, Tolerability, and Efficacy of ISV-303 to DuraSite Vehicle in Cataract Surgery Subjects
Brief Title: Comparison Study of ISV-303 to DuraSite Vehicle in Cataract Surgery Subjects
Acronym: ISV-303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-11-303-003
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Ocular Inflammation
MeSH Terms: interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ISV-303 (Experimental): 0.075% bromfenac in DuraSite vehicle dosed BID
  Interventions: Drug: ISV-303
- DuraSite Vehicle (Placebo Comparator): DuraSite Vehicle dosed BID
  Interventions: Other: DuraSite Vehicle

INTERVENTIONS:
Drug: ISV-303 — Bromfenac in DuraSite
  Arms: ISV-303
Other: DuraSite Vehicle — DuraSite Vehicle
  Arms: DuraSite Vehicle

SUMMARY:
The purpose of this study is to evaluate the ocular safety, tolerability, and efficacy of topical administration of ISV-303 compared with DuraSite Vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 or older scheduled for unilateral cataract surgery with posterior chamber intraocular lens implantation
* If a female is of childbearing potential, the subject must agree to and submit a negative pregnancy test before any protocol-specific procedures are conducted. The subject must use effective contraception for the duration of the study. Post menopausal is defined as having no menses for at least 12 consecutive months
* Signature of the subject on the Informed Consent Form
* Willing to avoid disallowed medication for the duration of the study.
* Willing and able to follow all instructions and attend all study visits
* Able to self-administer study drug (or have a caregiver available to instill all doses of study drug)
* Additional inclusion criteria also apply

Exclusion Criteria:

* Known hypersensitivity or poor tolerance to bromfenac sodium or any component of the study medications or any of the procedural medications
* Currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive pregnancy test
* Currently suffer from alcohol and/or drug abuse
* Prior (within 30 days of beginning study treatment) or anticipated concurrent use of an investigational drug or device
* A condition or a situation, which in the investigator's opinion may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation
* Additional exclusion criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- ISV-303: 0.075% bromfenac in DuraSite dosed BID
- Vehicle: DuraSite vehicle dosed BID
Period: Overall Study
Arm/Group | ISV-303 | Vehicle
Started | 180 | 88
Safety Population | 169 | 85
mITT Population | 168 | 85
Completed | 139 | 33
Not Completed | 41 | 55

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat: subjects who were randomized into the trial, underwent cataract surgery, and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-303 | Vehicle | Total
Number analyzed (Participants) | 168 | 85 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (10.14) | 68.4 (10.27) | 68.7 (10.17)
Age, Customized [Number; unit: participants]
  < 65 years | 47 | 25 | 72
  ≥ 65 years | 121 | 60 | 181
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 50 | 158
  Male | 60 | 35 | 95

OUTCOME MEASURES:

1. Primary Outcome: Ocular Inflammation
Description: Anterior chamber cell grade 0 at Day 15 measured on a 0 to 4 scale where "0" is 0 cells; "1" is 1-10 cells; "2" is 11-20 cells; "3" is 21-50 cells; "4" is > 50 cells, and no rescue medications.
Time Frame: 15 days
Population: Modified Intent-to-Treat (ITT) Population using Last Observation Carried Forward (LOCF) method.
Measure: Number; unit: participants
Arm/Group | ISV-303 | Vehicle
Number analyzed (Participants) | 168 | 85
participants | 96 | 16

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | ISV-303 | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/169 | 1/85
Other Adverse Events (participants affected / at risk) | 27/169 | 22/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-303 (N=169) | Vehicle (N=85)
Endophthalmitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-303 (N=169) | Vehicle (N=85)
Eye pain (Eye disorders) | 8 | 11
Iritis (Eye disorders) | 3 | 5
Ocular hypertension (Eye disorders) | 16 | 3
Headache (Nervous system disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other